CLINICAL TRIAL: NCT01941407
Title: A PHASE II TRIAL EVALUATING THE COMBINATION OF ERIBULIN (HALAVEN®) + BEVACIZUMAB (AVASTIN®) AS A FIRST LINE TREATMENT IN PATIENTS WITH METASTATIC HER2- BREAST CANCER
Brief Title: First Line Metastatic Breast Cancer Treatment (ESMERALDA)
Acronym: ESMERALDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-BR110
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Association eribulin and bevacizumab (Experimental): Drug: eribulin 1,23mg/m²; d1 and d8 in IV, all 3 weeks until 6 cycles or progression Drug: bevacizumab 15m/kg ; d1 in IV, all 3 weeks until 6 cycles or progression or toxicity
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — Eribulin: 1,23mg/m² d1, d8, IV Bevacizumab: 15mg/kg d1, IV
  Other Names: Drug: Bevacizumab

SUMMARY:
The efficacy of eribulin is now well known in metastatic breast cancer. Furthermore, a phase III combine study ( chemo + bev)in metastatic first line shown a gain in PFS with no extra toxicities.

It could be interesting to explore the combination of bev + eribulin in first line metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans
* Patient with metastatic mammary adenocarcinoma
* Hormone receptors ER and PR positive or negative for HER 2 negative

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Previous treatment with eribulin or bevacizumab
* Presence of symptomatic brain metastases or meningeal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of patient with non progressive disease | 12 months
  The principal endpoint is to determine the disease control rate (or rate of non-progression) at one year in patients with metastatic breast cancer treated in the first line setting by a combination of eribulin/bevacizumab.
  In this open-label trial, the sample size is calculated based on Simon's two-stage design, used to test whether the disease control rate at one year will be at least 50%, a clinically promising rate, versus a rate of 33%, a rate that is not clinically promising.
  Considering a type I risk (alpha) error of 5%, with 54 patients, this study has an 80% power to detect a disease control rate at one year of 50%.

SECONDARY OUTCOMES:
Toxicity based on the CTCAE v4.03 criteria | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire HARDY-BESSARD, MD, Principal Investigator — Clinique Armoricaine de Radiologie
Locations (40):
- France (40):
  - Centre Paul Papin, Angers
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Ste Catherine, Avignon
  - Clinique Tivoli, Bordeaux
  - Hôpital Fleyriat, Bourg-en-Bresse
  - Hôpital Morvan - Centre Hospitalier Universitaire, Brest
  - centre Francois baclesse, Caen
  - Hôpital Privé Sainte-Marie, Chalon-sur-Saône
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre d'Oncologie et de Radiothérapie, Dijon
  - Centre Hospitalier la Dracénie, Draguignan
  - Centre Hospitalier Intercommunal, Fréjus
  - Hôpital Privé Drôme Ardèche - Clinique Pasteur, Guilherand-Granges
  - Clinique de la Sauvegarde, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Clairval, Marseille
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - Centre d'oncologie de Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Régional, Orléans
  - Institut Curie - Hopital Claudius Régaud, Paris
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Saint-Joseph, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - Centre Hospitalier Lyon-sud, Pierre-Bénite
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - Clinique Courlancy, Reims
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Anne-Claire Hardy-Bessard, MD, Saint-Brieuc
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Centre Hospitalier Privé de Saint-Grégoire, Saint-Grégoire
  - GHPSO - Site Senlis, Senlis
  - Centre de Radiothérapie - Clinique Sainte-Anne, Strasbourg
  - Centre Hospitalier de Thonon-les-Bains, Thonon-les-Bains
  - Clinique Pasteur, Toulouse
  - CHU Bretonneau, Tours
  - Centre Hospitalier de Valence, Valence
  - Centre Hospitalier Bretagne Atlantique, Vannes